CLINICAL TRIAL: NCT02957786
Title: RAUORA: Cytisine Versus Varenicline for Smoking Cessation
Brief Title: Cytisine Versus Varenicline for Smoking Cessation
Acronym: RAUORA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Lakes District Health Board (Other); Brunel University (Other)
Responsible Party: Principal Investigator, Natalie Walker, Associate Professor, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTN: U1111-1187-2838
Record Dates: First submitted 2016-10-27; First posted 2016-11-08 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Smoking Cessation
Keywords: cytisine; varenicline; smoking cessation; indigenous
MeSH Terms: conditions — Smoking Cessation | interventions — cytisine; Varenicline

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cytisine plus behavioural support (Experimental): 12-week course of cytisine capsules (1.5mg), with a decreasing dosing regimen (9mg/day for days 1-3, 7.5mg/day for days 4-12, 6mg/day for days 13-16, 4.5mg/day for days 17-20, 3.0mg/day from days 21-week 12).
  Participants will be asked to reduce their smoking over the first four days of treatment so that they are not smoking at all by the fifth day, which will be their designated Quit date.
  Participants will also withdrawal-orientated behavioural support (delivered by cessation advisors), in addition to brief cessation advice from the study-specific doctor (at the point that the prescription is provided) and community pharmacist (at the point the participant redeems their prescription).
  Interventions: Drug: Cytisine; Behavioral: Behavioural support
- Varenicline plus behavioural support (Active Comparator): 12-week course of Varenicline tablets (0.5mg/1mg), with an increasing dosing regimen (0.5mg/day for days 1-3, 1.0mg/day for days 4-7, 2.0mg/day for day 8-week 12).
  Participants will be asked to reduce their smoking over the first four days of treatment so that they are not smoking at all by the fifth day, which will be their designated Quit date.
  Participants will also receive withdrawal-orientated behavioural support (delivered by cessation advisors), in addition to brief cessation advice from the study-specific doctor (at the point that the prescription is provided) and community pharmacist (at the point the participant redeems their prescription).
  Interventions: Behavioral: Behavioural support; Drug: Varenicline

INTERVENTIONS:
Drug: Cytisine — Cytisine tablets
  Other Names: Tabex
  Arms: Cytisine plus behavioural support
Behavioral: Behavioural support — Withdrawal-orientated cessation support
Drug: Varenicline — Varenicline tablets
  Other Names: Champix
  Arms: Varenicline plus behavioural support

SUMMARY:
To evaluate the effectiveness, safety, and cost-effectiveness of cytisine plus behavioural support compared to varenicline plus behavioural support for smoking cessation, in indigenous Māori (or family of Māori) who smoke and are motivated to quit.

DETAILED DESCRIPTION:
Cytisine, a natural product, found in plants such as the Golden Rain and New Zealand Kowhai, partially blocks the effects of nicotine on the brain. Cytisine has been used as a smoking cessation treatment in several Central and Eastern European countries since the 1960s, is inexpensive compared to other cessation medications and has few known side effects. New Zealand research has shown cytisine to be more effective than nicotine replacement therapy at helping people quit smoking. Using a clinical trial design (N=2140) the investigators plan to investigate whether cytisine is at least as good as varenicline (the most effective, but most expensive, smoking cessation medication currently available in New Zealand) for helping Māori/family of Māori who smoke, to quit.

ELIGIBILITY:
Inclusion Criteria:

* daily tobacco smokers
* self-identify as Māori (indigenous New Zealander) or whānau (family) of Māori
* want to stop smoking in the next two weeks
* are at least 18 years of age
* are able to provide verbal consent
* reside in the Lakes District Health Board, Eastern Bay of Plenty or Tokoroa region at the time of enrolment
* have daily access to a mobile phone with text capability and/or email and access to the internet via computer or smartphone
* are eligible for subsidised varenicline under special authority conditions

Exclusion Criteria:

* are pregnant or breastfeeding
* are current users of other smoking cessation therapies (e.g. nicotine replacement therapy [NRT], buproprion [Zyban], clonidine, nortriptyline, e-cigarettes)
* are enrolled in another smoking cessation programme or another smoking cessation study
* have a contraindication for cytisine or varenicline
* have used varenicline or cytisine in the past 12 months
* have another person in their household involved in the trial
* have moderate or severe renal impairment,
* are being treated for active or latent TB
* have been treated for a heart attack, stroke, or severe angina within the last two weeks
* have uncontrolled high blood pressure (> 150 mmHg systolic, > 100 mmHg diastolic)
* have a history of seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 679 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Continuous abstinence from smoking | Six months post-quit date
  Self-report of smoking not more than five cigarettes from the quit date, supported by biochemical validation using a carbon monoxide (CO) expired breath

SECONDARY OUTCOMES:
Continuous abstinence from smoking | One month post-quit date
  Self-report of smoking not more than five cigarettes from the quit date
Continuous abstinence from smoking | Three months post-quit date
  Self-report of smoking not more than five cigarettes from the quit date
Continuous abstinence from smoking | 12 months post-quit date (in 2/3 of sample)
  Self-report of smoking not more than five cigarettes from the quit date, supported by biochemical validation using a carbon monoxide (CO) expired breath
7-day point prevalence abstinence from smoking | One month post-quit date
  Self-report of having smoked no cigarettes (not even a puff) in the past seven days.
7-day point prevalence abstinence from smoking | Three month post-quit date
  Self-report of having smoked no cigarettes (not even a puff) in the past seven days.
7-day point prevalence abstinence from smoking | Six month post-quit date
  Self-report of having smoked no cigarettes (not even a puff) in the past seven days,supported by biochemical validation using a carbon monoxide (CO) expired breath.
7-day point prevalence abstinence from smoking | 12 month post-quit date (in 2/3 of sample)
  Self-report of having smoked no cigarettes (not even a puff) in the past seven days,supported by biochemical validation using a carbon monoxide (CO) expired breath.
Time to relapse back to smoking | One month post-quit date
  Defined as return to daily smoking.
Time to relapse back to smoking | Three month post-quit date
  Defined as return to daily smoking.
Time to relapse back to smoking | Six month post-quit date
  Defined as return to daily smoking.
Time to relapse back to smoking | 12 month post-quit date (in 2/3 of sample)
  Defined as return to daily smoking.
Cigarette withdrawal | One month post-quit date
  The physical signs and symptoms associated with nicotine withdrawal over the last week, measured using the Mood and Physical Symptoms Scale (MPSS)
Cigarette withdrawal | Three months post-quit date
  The physical signs and symptoms associated with nicotine withdrawal over the last week, measured using the Mood and Physical Symptoms Scale (MPSS)
Cigarette withdrawal | Six months post-quit date
  The physical signs and symptoms associated with nicotine withdrawal over the last week, measured using the Mood and Physical Symptoms Scale (MPSS)
Cigarettes per day | One month post-quit date
  Number of cigarettes smoked per day, if smoking
Cigarettes per day | Three month post-quit date
  Number of cigarettes smoked per day, if smoking
Cigarettes per day | Six month post-quit date
  Number of cigarettes smoked per day, if smoking
Cigarettes per day | 12 month post-quit date (in 2/3 of sample)
  Number of cigarettes smoked per day, if smoking
Smoking satisfaction, if smoking | One month post-quit date
  Measured using the modified Cigarette Evaluation Questionnaire (mCEQ).
Smoking satisfaction, if smoking | Three month post-quit date
  Measured using the modified Cigarette Evaluation Questionnaire (mCEQ).
Smoking satisfaction, if smoking | Six month post-quit date
  Measured using the modified Cigarette Evaluation Questionnaire (mCEQ).
Health-related quality of life | One month post-quit date
  Measured using the New Zealand EQ-5D Tariff 2
Health-related quality of life | Three months post-quit date
  Measured using the New Zealand EQ-5D Tariff 2
Health-related quality of life | Six months post-quit date
  Measured using the New Zealand EQ-5D Tariff 2
Acceptability of allocated treatment | One month post-quit date
  Participants will be asked for their views on the use of their allocated medication as a cessation aid (i.e. whether they would recommend the treatment to another smoker and the things they liked or disliked about using the product).
Acceptability of allocated treatment | Three months post-quit date
  Participants will be asked for their views on the use of their allocated medication as a cessation aid (i.e. whether they would recommend the treatment to another smoker and the things they liked or disliked about using the product).
Use of other methods of cessation | One month post-quit date
  Participants will be asked about their use of other methods of cessation, such as NRT, Zyban, clonidine, nortriptyline, e-cigarettes, acupuncture etc.
Use of other methods of cessation | Three months post-quit date
  Participants will be asked about their use of other methods of cessation, such as NRT, Zyban, clonidine, nortriptyline, e-cigarettes, acupuncture etc.
Use of other methods of cessation | Six months post-quit date
  Participants will be asked about their use of other methods of cessation, such as NRT, Zyban, clonidine, nortriptyline, e-cigarettes, acupuncture etc.
Medication compliance | One month post-quit date
  Self-reported pill count, early stopping of allocated medication and reasons why.
Medication compliance | Three months post-quit date
  Self-reported pill count, early stopping of allocated medication and reasons why.
Adverse events | One month post-quit date
  Any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study treatment, whether or not it is considered related to the product.
Adverse events | Three month post-quit date
  Any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study treatment, whether or not it is considered related to the product.
Adverse events | Six month post-quit date
  Any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study treatment, whether or not it is considered related to the product.
Adverse events | 12 month post-quit date (in 2/3 of sample)
  Any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study treatment, whether or not it is considered related to the product.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Walker, PhD, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- National Institute for Health Innovation, University of Auckland, Auckland, North Island, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
IPD analysis planned - details of plan not yet finalized

REFERENCES:
- [Background] Walker N, Smith B, Barnes J, Verbiest M, Kurdziel T, Parag V, Pokhrel S, Bullen C. Cytisine versus varenicline for smoking cessation for Maori (the indigenous people of New Zealand) and their extended family: protocol for a randomized non-inferiority trial. Addiction. 2019 Feb;114(2):344-352. doi: 10.1111/add.14449. Epub 2018 Nov 9. PMID 30276931
- [Result] Walker N, Smith B, Barnes J, Verbiest M, Parag V, Pokhrel S, Wharakura MK, Lees T, Cubillos Gutierrez H, Jones B, Bullen C. Cytisine versus varenicline for smoking cessation in New Zealand indigenous Maori: a randomized controlled trial. Addiction. 2021 Oct;116(10):2847-2858. doi: 10.1111/add.15489. Epub 2021 May 4. PMID 33761149